CLINICAL TRIAL: NCT03456856
Title: Open-label, Single-arm, Study Assessing the Efficacy and Safety of Ivabradine (Corlanor) in African-American/Black Subjects With Heart Failure and Left Ventricular Systolic Dysfunction
Brief Title: A Study of Ivabradine in African-American/ Black Subjects With Heart Failure and Left Ventricular Systolic Dysfunction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160231
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure (HF)
Keywords: Cardiac; Congestive; Decompensation; Heart Failure; Left-Sided; Myocardial; Corlanor; Ivabradine; African American; Black; Michigan
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivabradine (Experimental): The starting dose of ivabradine was 5 mg twice daily (BID), although investigators had the discretion to start participants at 2.5 mg BID if participant had a history of conduction defects, or bradycardia that could lead to hemodynamic compromise. Dose was adjusted at Day 15 (and at any other clinical visit) between 2.5 - 7.5 mg BID based on heart rate and signs/symptoms of bradycardia.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Film-coated tablets taken orally with food twice a day. Tablets supplied in strengths of 5.0 mg and 7.5 mg. 5.0 tablets were split into equal halves for dosages of 2.5 mg.
  Other Names: Corlanor®

SUMMARY:
This study is a prospective, open-label, single-arm intervention study in African-American/Black subjects with heart failure and reduced ejection fraction (HFrEF).

There will be a 7-day screening period, a 57-day open-label treatment period, and a safety follow-up at day 87 or 30 days after the last administration of the investigational product.

DETAILED DESCRIPTION:
The goal of this study is to determine the impact of adding ivabradine therapy to the standard of care (SOC) in African-American/Black subjects with Heart Failure (HF) and reduced ejection fraction (HFrEF) on changes in heart rate (HR) from baseline (SOC alone). Changes in HR from baseline will be correlated with the changes from baseline in activity level of the subjects, as measured by both a standard 6-minute walk distance and an accelerometer device.

The primary hypothesis is that ivabradine effectively reduces HR between baseline and day 57 in African-American/Black subjects. Because mean reductions of approximately 5 beat per minute (bpm) have been observed in the overall placebo-treated subjects in the SHIFT study as well as in the placebo-treated subjects of the subgroup analysis of non-African-American/Black subjects enrolled in the SHIFT study, we will test whether the mean reduction with ivabradine exceeds 5 bpm, and estimate the degree to which the mean reduction with ivabradine exceeds 5 bpm.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any study specific activities/ procedures
* Male or female subject ≥ 18 years of age, describing self as African American/Black
* Must have a diagnosis of heart failure (HF) confirmed by medical records, be in stable condition, and treated with stable optimal pharmacological therapy as per their personal physician's care.
* Left ventricular ejection fraction (LVEF) ≤ 35% confirmed by investigator
* New York Heart Association (NYHA) class II to IV assessed at the time of screening
* Electrocardiogram (ECG) documentation at the time of screening of sinus rhythm with resting heart rate (HR) ≥ 70 bpm by local ECG reading
* Must be able to complete a 6-minute walk test (6MWT) and wear an accelerometer

Exclusion Criteria:

* Recent myocardial infarction (≤ 2 months) or stroke (≤ 1 month) prior to enrollment
* If the subject received within 3 months before or is scheduled to receive within 42 days after enrollment any of the following: revascularization, ventricular assist device, continuous or intermittent inotropic therapy, hospice care, major organ transplant, or is receiving renal replacement therapy by dialysis
* If the subject received implantation of a cardioverter defibrillator or cardiac resynchronization therapy within 42 days before or is scheduled to receive implantation of a cardioverter defibrillator or cardiac resynchronization therapy within 42 days after enrollment
* Severe primary valve disease or scheduled for surgery for valvular heart disease
* Pacemaker with atrial or ventricular pacing (except bi-ventricular pacing) >40% of the time, or with a stimulation threshold at the atrial or ventricular level ≥ 60 bpm
* Permanent atrial fibrillation or flutter
* Sick sinus syndrome, sinoatrial block, or second and third degree atrio-ventricular block
* History of symptomatic or sustained (≥ 30 sec) ventricular arrhythmia unless a cardioverter defibrillator was implanted
* History of congenital QT syndrome
* Any cardioverter defibrillator shock experienced within 1 month of enrollment
* Hypertrophic obstructive cardiomyopathy, active myocarditis or constrictive pericarditis, or clinically significant congenital heart disease
* Chronic antiarrhythmic therapy (except digitalis)
* Scheduled outpatient intravenous (IV) infusions for HF (eg, inotropes,vasodilators [eg, nesiritide], diuretics) or routinely scheduled ultrafiltration
* Evidence of digitalis intoxication within 7 days prior to screening
* Systolic blood pressure > 180 mm Hg or < 90 mm Hg, or diastolic blood pressure > 110 mm Hg or < 50 mm Hg at any time during the screening phase
* Known untreated hypothyroidism or hyperthyroidism, adrenal insufficiency, active vasculitis due to collagen vascular disease
* Have known acute or serious co-morbid condition (e.g, major infection or hematologic, renal, hepatic, metabolic, gastrointestinal or endocrine dysfunction) that may interfere with the study, or severe concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 1 year or malignancy within 5 years prior to enrollment with the following exceptions: localized basal or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia
* Subjects taking QT prolonging medicinal products for cardiovascular (e.g, but not limited to, quinidine, disopyramide, bepridil, sotalol, ibutilide, amiodarone) or non-cardiovascular disease (e.g, but not limited to, pimozide, ziprasidone, sertindole, mefloquine, halofantrine, pentamidine, cisapride, IV erythromycin).
* Subjects exposed to a strong CYP3A4 inhibitor (examples of strong CYP3A4 inhibitors include; azole antifungals [eg, itraconazole], macrolide antibiotics [e.g, clarithromycin, telithromycin], human immunodeficiency virus (HIV) protease inhibitors, [eg, nelfinavir], and nefazodone]) within 14 days prior to enrollment, or to a strong CYP3A4 inducer (examples of CYP3A4 inducers include; St. John's wort, rifampicin, barbiturates, and phenytoin) within 28 days prior to enrollment
* Subjects who received diltiazem or verapamil within 48 hours prior to enrollment.
* Previously received ivabradine prior to participation in this study
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 14 days after the last dose of investigational product. Females of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive urine pregnancy test.
* Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 14 days after the last dose of investigational product.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject likely not to be available to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Wilmington, Delaware
  - Research Site, Detroit, Michigan
  - Research Site, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Lanfear DE, Neaton KR, Lu C, Liu Y, Dent-Acosta RE. A Phase 4, Open-Label, Single-Arm Study Assessing the Efficacy and Safety of Ivabradine in African American Patients with Heart Failure and Reduced Ejection Fraction. Cardiol Ther. 2020 Dec;9(2):561-568. doi: 10.1007/s40119-020-00196-1. Epub 2020 Aug 17. PMID 32808163
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 participants were enrolled at 2 centers in the United States.
Period: Overall Study
Arm/Group | Ivabradine
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set which included all enrolled participants.
Arm/Group | Ivabradine
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.6)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 24
  65-74 years | 5
  75-84 years | 0
  >=85 years | 1
  Unknown | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — NYHA Classification
  * Class I-No symptoms and no limitation in ordinary physical activity
  * Class II-Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  * Class III-Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 meters). Comfortable only at rest.
  * Class IV-Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  * No NYHA class listed or unable to determine.
  Participants
    NYHA Class I | 0
    NYHA Class II | 22
    NYHA Class III | 8
    NYHA Class IV | 0
Primary Cause of Heart Failure [Count of Participants; unit: Participants]
  Ischemic heart disease | 5
  Non-ischemic heart disease | 25
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage total blood in left ventricle] — Left ventricular ejection fraction (LVEF) is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. A normal left ventricular ejection fraction (LVEF) ranges from 55% to 70%. LVEF was measured by echocardiogram.
  percentage total blood in left ventricle | 25.6 (6.8)
Baseline Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Baseline was defined as the last no-missing value collected prior to or on Study Day 1.
  Heart rate was measured by 12-lead ECG.
  beats per minute | 83.6 (8.9)
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Baseline was defined as the last non-missing value collected prior to or on Study Day 1.
  mmHg | 126.8 (17.1)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Baseline was defined as the last non-missing value collected prior to or on Study Day 1.
  mmHg | 73.0 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Heart Rate (HR) at Day 57
Description: Summary is based on observed data, and no imputation is used for missing values.
  Least-square mean is from the repeated measures model which includes scheduled visits and baseline HR measurement as covariates.
  The mean change from baseline in heart rate is compared to -5 beats/min which is observed in the placebo group in the Systolic Heart Failure Treatment with the IF Inhibitor Ivabradine Trial (SHIFT) study ( NCT02441218, PMID 20801500).
Time Frame: Day1 (baseline), Day 57
Population: Full analysis set which included all enrolled participants.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Ivabradine
Number analyzed (Participants) | 30
beats per minute | -9.5 (1.7)
Statistical Analysis 1: Comparison: Ivabradine; The estimated mean treatment difference (95% CI) takes into account a presumed -5 bpm change from baseline heart rate in the absence of ivabradine (as seen in the placebo group in the SHIFT study, (NCT02441218, PMID 20801500); Test type: Superiority; p = 0.013, repeated measures linear model; least square mean difference = -4.5, 95% CI 2-sided [-8.0 to -1.0], Standard Error of Mean 1.7

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 87 (30 days after the last dose of IP)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Ivabradine
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivabradine (N=30)
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ivabradine (N=30)
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03456856/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03456856/SAP_001.pdf